CLINICAL TRIAL: NCT01584947
Title: Clinical Trials With a Local Anesthetic Lozenge for the Treatment of Oral Mucosal Pain in Burning Mouth Syndrome, Sjögrens Syndrome and Lichen Planus.
Brief Title: Clinical Trials With a Local Anesthetic Lozenge for the Treatment of Chronic Oral Pain
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Because of a very slow patient recruitment.
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Oracain II Aps (Unknown)
Responsible Party: Principal Investigator, Anne Marie Lynge Pedersen, Dentist, PhD, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2011-006196-19
Record Dates: First submitted 2012-04-23; First posted 2012-04-25 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Chronic Pain
Keywords: Oral pain; Local anesthetic; Bupivacaine hydrochloride
MeSH Terms: conditions — Chronic Pain | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo lozenge (Placebo Comparator): The patients will be randomized to start two weeks treatment with either a bupivacaine lozenge or a placebo lozenge (taken three times a day). The two weeks treatment is followed by a week without treatment. Afterwards they start another two weeks treatment with the opposite type of lozenge from the first treatment period.
  Interventions: Drug: Placebo
- Bupivacaine lozenge (Active Comparator): The patient will be randomized to start two weeks treatment with either a bupivacaine lozenge or a placebo lozenge (taken three times a day). The two weeks treatment is followed by a week without treatment. Afterwards the patient starts another two weeks treatment with the opposite type of lozenge from the first treatment period.
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine — Bupivacaine lozenge taken 3 times a day for two weeks
  Arms: Bupivacaine lozenge
Drug: Placebo — Placebo lozenge taken three times a day for two weeks
  Arms: Placebo lozenge

SUMMARY:
The aim of the project is to do a fase two trial, where the effect of a local anesthetic lozenge will be tested in regard to oral pain, dryness of the mouth, irregularity of taste as well as investigate a potential antiinflammatory effect in patients with burning mouth syndrome, Sjögrens syndrome and lichen planus.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with burning mouth syndrome, Sjögrens syndrome or lichen planus
* All fertile women need to use save contraception
* Age between 18 and 75 years
* Able to speak, read and understand the danish language
* Must be informed orally and release a written consent and a signed authorization statement

Exclusion Criteria:

* Pregnant or breastfeeding women
* Known allergy to bupivacaine or other local anesthetics of the amide type
* Active infection which requires antibiotic treatment
* Patients in immune suppressive treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2012-04; Primary Completion 2014-01 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Assessment of oral pain on the Visual Analog Scale | The patients assess their oral pain when they attend the four examinations and they fill in a diary for a total of four weeks.
  Assessment of oral pain in patients with burning mouth syndrome, Sjögrens syndrome or lichen planus after treatment with a bupivacaine lozenge or a placebo lozenge.
  The patient assess their oral pain on the visual analog scale when they attend the four examinations. The patients also fill in a diary for a total of four weeks where they are in treatment where they assess VAS for pain, dryness of the mouth and irregularity of taste

SECONDARY OUTCOMES:
Measure the inflammation markers in blood, saliva and tissue | Blood- and saliva samples are taken the four times the patient attend the examinations. They are taken over a periode of five weeks. Tissue samples are taken before the first treatment period starts and when the final treatment period is finished.
  The inflammation markers in blood, saliva and tissue will be analyzed to investigate if there are changes in the level in patients with chronic oral pain.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Marie L Pedersen, Ph.d., Principal Investigator — Department of Odontology, University of Copenhagen
Locations (1):
- Department of Odontology, University of Copenhagen, Copenhagen, Denmark